CLINICAL TRIAL: NCT00172068
Title: Efficacy and Tolerability of Intravenous Zometa® (Zoledronic Acid) 4 mg in Primary Breast Cancer Patients With Disseminated Tumor Cells in Bone Marrow. A Prospective, Randomized, Parallel Group, Open-label, Clinical Pilot Study.
Brief Title: Zoledronic Acid in the Treatment of Breast Cancer With Minimal Residual Disease in the Bone Marrow
Acronym: MRD-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446GDE05
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Primary Breast Cancer
Keywords: Primary breast cancer; Bone metastases; Minimal residual disease; Bisphosphonates
MeSH Terms: conditions — Neoplasm, Residual | interventions — Zoledronic Acid; Calcium; Vitamin D

ARMS (2):
- Treatment Group (Experimental)
  Interventions: Drug: Zoledronic acid + Calcium/Vitamin D
- Control Group (Active Comparator)
  Interventions: Drug: Zoledronic acid + Calcium/Vitamin D

INTERVENTIONS:
Drug: Zoledronic acid + Calcium/Vitamin D

SUMMARY:
Metastatic bone disease is an important prognostic factor for survival which will in median be close to two years after first diagnosis of osseous metastases. This open-label study will investigate the safety and efficacy of zoledronic acid in patients with breast cancer and minimal residual disease in the bone marrow.

ELIGIBILITY:
Inclusion Criteria:

* Patients, with primary breast cancer who had undergone complete primary tumor resection and axillary lymph node dissection
* Evidence of minimal residual disease (disseminated tumor cells in bone marrow)
* Patients had to receive one of the following adjuvant therapy categories: chemotherapy ± hormonal therapy or hormonal therapy alone

Exclusion Criteria:

* Inflammatory, metastatic or recurrent breast cancer or a history of breast cancer prior to the currently diagnosed case
* Neo-adjuvant chemotherapy, neo-adjuvant hormonal therapy, or neo-adjuvant radiotherapy
* Prior stem cell rescue/bone marrow transplant
* History of other cancers aside from non-melanomatous skin cancer or carcinoma in situ of the uterine cervix

Additional protocol-defined inclusion / exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2002-01; Primary Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Reduction of detected tumor cells in bone marrow | 12 months

SECONDARY OUTCOMES:
Tumor cell detection in bone marrow in comparison to the time point of primary surgery (Baseline). | 24 months
Bone metastases-free survival | 24 months
Disease-free survival | 24 months
Bone mineral density | at 12 and 24 months
Number and localization of bone metastases | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (4):
- Germany (4):
  - Novartis Invstigative Site, Bielefeld
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Tübingen

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- [Derived] Banys M, Solomayer EF, Gebauer G, Janni W, Krawczyk N, Lueck HJ, Becker S, Huober J, Kraemer B, Wackwitz B, Hirnle P, Wallwiener D, Fehm T. Influence of zoledronic acid on disseminated tumor cells in bone marrow and survival: results of a prospective clinical trial. BMC Cancer. 2013 Oct 15;13:480. doi: 10.1186/1471-2407-13-480. PMID 24128322